CLINICAL TRIAL: NCT07202377
Title: Impact of Real-time MIC (Minimum Inhibitory Concentration) Reporting (<6 Hours) on β-lactam Prescription in Cases of Gram-negative Bacilli Bacteremia in ICU Patients in Real-life Settings
Acronym: CMIBActRéa
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP240793
Record Dates: First submitted 2025-08-22; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Gram-negative Bacteremia; Intensive Care Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Performance of an antibiotic susceptibility test on agar medium (Active Comparator): Performance of an antibiotic susceptibility test on agar medium, with results expected between H18 and H24
  Interventions: Diagnostic Test: antibiotic susceptibility testing on agar medium
- Antibiotic susceptibility testing performed using the Reveal technique (Experimental): Antibiotic susceptibility testing performed using the Reveal technique, with results available between the 4th and 6th hour (H4-H6) after blood culture positivity, allowing for rapid clinical categorization for the 23 antibiotics tested, along with their corresponding MICs.
  Interventions: Diagnostic Test: SPECIFIC REVEAL® Rapid AST system

INTERVENTIONS:
Diagnostic Test: SPECIFIC REVEAL® Rapid AST system — The SPECIFIC REVEAL™ system uses biosensors capable of detecting volatile substances released by microorganisms during their growth. The detection of these volatile compounds by ultra-high-performance biosensors enables very early detection of bacterial growth compared with standard technologies based on visual systems (e.g. diffusion antibiogram or MICs determined by microdilution in liquid media) or optical density measurement systems (e.g. Vitek2)
  Arms: Antibiotic susceptibility testing performed using the Reveal technique
Diagnostic Test: antibiotic susceptibility testing on agar medium — Performance of an antibiotic susceptibility test on agar medium, with results expected between H18 and H24
  Arms: Performance of an antibiotic susceptibility test on agar medium

SUMMARY:
Evaluate the impact of rapid, real-time (4 to 6 h) MIC reporting compared with the standard method (=diffusion antibiotic susceptibility testing) (18 to 24 h) on β-lactam prescribing in terms of the choice of molecule by the resuscitating clinician in the event of real-life Gram-negative Bacilli GNB bacteremia in the ICU.

DETAILED DESCRIPTION:
In the microbiology laboratory, antibiotic susceptibility is traditionally determined using the disk diffusion method on agar medium, directly from a positive blood culture bottle, which requires 18 to 24 hours of incubation. Over the past decade, the turnaround time for antibiotic susceptibility testing has been shortened (down to 7 hours) thanks to rapid diagnostic tools. However, to date, there is no rapid (within 4 to 6 hours) and accurate method for determining the Minimum Inhibitory Concentration (MIC) that would allow for optimized antibiotic treatment beyond the basic susceptibility to a tested drug. This level of precision would be particularly useful in critically ill septic patients, especially in cases of bacteremia caused by Gram-negative bacilli (GNB).

Recent intensive care guidelines have suggested that for β-lactam antibiotics, the therapeutic target in these patients should be a plasma antibiotic concentration between 4 to 8 times the MIC of the administered antibiotic, depending on the bacterium and the drug. MIC thus represents a key determinant for optimizing antibiotic therapy by increasing the likelihood of achieving the pharmacodynamic efficacy targets of β-lactams.

The use of a new instrument, the SPECIFIC REVEAL® Rapid AST system (bioMérieux), which provides not only a full antibiogram but also MIC values for 23 different antibiotics as early as 4 hours after a positive GNB blood culture (Enterobacterales, Pseudomonas aeruginosa, Acinetobacter baumannii), could represent a potential benefit for ICU patients by enabling rapid optimization of antibiotic therapy. This technique was validated by comparison with two reference methods: a precise MIC determination method (broth microdilution, Sensititre, ThermoFisher) and an approximate method (Vitek2, bioMérieux). A 96% correlation was observed across the 23 antibiotics tested. Furthermore, a recent study conducted outside the ICU suggested a clinical impact, with earlier re-evaluation of antibiotic choices in 58% of cases.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged over 18 years
* Patients with a positive blood culture for Gram-negative bacilli (Enterobacterales, Pseudomonas aeruginosa, Acinetobacter baumannii) with results reported on weekdays before 11:00 ante meridiem (AM)
* Patients clinically suspected of infection
* Treated with empirical antibiotic therapy including a β-lactam, among the standard list of antibiotics to be tested recommended by CASFM-EUCAST (European Committee on Antimicrobial Susceptibility Testing) for Enterobacterales/Pseudomonas and included in the Reveal Rapid AST System panel
* Hospitalized in intensive care unit (ICU) for at least the next 24 hours
* Written informed consent obtained from the patient or a relative for study participation (emergency consent)
* Affiliated with the French social security system

Exclusion Criteria:

* Patients receiving withdrawal or limitation of care
* Patients with an expected survival prognosis of less than 72 hours
* Patients with bloodstream infections caused by Gram-negative bacilli other than Acinetobacter baumannii, Citrobacter freundii, Citrobacter koseri, Enterobacter cloacae, Escherichia coli, Klebsiella aerogenes, Klebsiella oxytoca, Klebsiella pneumoniae, Proteus mirabilis, or Pseudomonas aeruginosa
* Patients treated with antibiotic therapy not including a β-lactam
* Polymicrobial bloodstream infections
* Pregnant or breastfeeding women
* Patients under legal protection (guardianship or conservatorship)
* Participation in another interventional research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients for whom antibiotic therapy was modified in terms of molecule selection within the first 24 hours following the report of a positive blood culture for Gram-negative bacilli, based on medical prescriptions after inclusion | 24 hours following the report of a positive blood culture for Gram-negative bacilli
  To evaluate whether the rapid and real-time reporting (4 to 6 hours) of MICs, compared to the standard method (i.e., disk diffusion antibiogram, 18 to 24 hours), has an impact on β-lactam prescription in terms of molecule selection by the ICU clinician in real-life cases of bloodstream infections due to Gram-negative bacilli.

SECONDARY OUTCOMES:
Proportion of patients with favorable clinical and biological evolution based on the Sequential Organ Failure Assessment (SOFA) score between H72 and H96, and on day 7 | hour72 and hour96, and on day 7
  To evaluate the impact of rapid MIC reporting compared to the standard method (i.e., disk diffusion, which provides only clinical categorization) on clinical and biological outcomes between H72 and H96, and on day 7
Proportion of patients with favorable microbiological evolution, defined by negative blood cultures collected between H72 and H96. | hour72 and hour96
  To evaluate the impact of rapid MIC reporting compared to the standard method (i.e., disk diffusion, which provides only clinical categorization) on microbiological evolution between H72 and H96
Plasma concentration/MIC ratio observed at the first β-lactam level measurement between H24 and H48 | hour24 and hour48
  To evaluate the impact of rapid MIC reporting compared to the standard method (i.e., disk diffusion, which provides only clinical categorization) on the probability of achieving a residual β-lactam plasma concentration between 4 and 8 times the MIC at the first antibiotic measurement between 24 and 48 hours (H24-H48).
Proportion of patients alive at day 30 (D30) and at ICU discharge | day 30
  To evaluate the impact of rapid MIC reporting compared to the standard method (i.e., disk diffusion, which provides only clinical categorization) on mortality at day 30 (D30) and at ICU discharge
Incidence of antibiotic-associated adverse events affecting renal, neurological, and hepatic function during the course of treatment | day 30
  To evaluate the impact of rapid MIC reporting compared to the standard method (i.e., disk diffusion, which provides only clinical categorization) on the incidence of antibiotic-related adverse effects (renal, neurological, hepatic tolerance) throughout the treatment.
Costs associated with rapid MIC testing, hospital stay, antibiotics, and microbiological tests as well as costs assessed at 30 days. | day 30
  To evaluate the medico-economic impact of the rapid MIC reporting strategy through a cost-consequence analysis, which allows for a disaggregated presentation of the consequences of rapid MIC reporting for patients, prescribers, and the microbiology department; costs are estimated from the healthcare provider's perspective